CLINICAL TRIAL: NCT06149013
Title: Efficacy of MindAhead's Digital Behavioral Activation Therapy in Adults with Mild Cognitive Impairment or Mild Dementia: a Monocentric Randomized Controlled Pilot Trial (MindMoments-Pilot)
Brief Title: Efficacy of MindAhead's Digital Behavioral Activation Therapy in Adults with MCI or Mild Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MindAhead UG (Industry)
Collaborators: University Medical Center Göttingen (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MiMo-P
Record Dates: First submitted 2023-11-09; First posted 2023-11-28 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Mild Cognitive Impairment; Mild Dementia
Keywords: Behavioral Activation Therapy; Active lifestyle intervention
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MindAhead + TAU Group (Experimental): The intervention group receives the digital health app MindAhead Active for 3 months as well as treatment-as-usual (TAU, see Control intervention).
  Interventions: Device: MindAhead Active; Other: Treatment-as-usual
- TAU Group (Active Comparator): The control group receives TAU which may include antidementive medication (e.g., acetylcholinesterase inhibitors), advice on protective lifestyle factors, vitamin supplementation, ergotherapy, cognitive training (including digital health apps), or statins depending on clinical findings.
  Interventions: Other: Treatment-as-usual

INTERVENTIONS:
Device: MindAhead Active — MindAhead's Active app focuses on increasing meaningful and enjoyable cognitive, physical, and social activities specifically adapted to patients with early cognitive decline (MCI or mild dementia). These techniques include psychoeducation (explaining the rationale, the components of behavioral activation, and protective activities), action planning (selecting activities, goal setting, activity scheduling, graded task assignment, written schedules, and step-by-step sequencing) and action/self-monitoring (assessing execution of and enjoyment in activities, monitor mood and cognitive problems), as well as value-based activation (understanding most important values, selecting activities according to these values). This process aims to enable the users to understand which activities are enjoyable and meaningful to them and how to implement these activities into their daily lives. MindAhead's Active app consists of one to five sessions per week.
  Other Names: MindAhead's Behavioral Activation Therapy
  Arms: MindAhead + TAU Group
Other: Treatment-as-usual — Depending on patient-specific clinical findings it includes antidementive medication (e.g., acetylcholinesterase inhibitors), advice on protective lifestyle factors, vitamin supplementation, ergotherapy, cognitive training (including digital health apps), or statins.
  Other Names: TAU

SUMMARY:
This pilot study investigates effects of a digital behavioral activation therapy in treating patients with mild cognitive impairment and mild dementia, applying a randomized controlled parallel group design. The primary goal is to estimate effect sizes for a larger trial. A further aim is to investigate the feasibility of study procedures and to validate new questionnaire scores. Primary outcomes are the change in the patients' quality of life and in their overall activity level.

DETAILED DESCRIPTION:
Face-to-face behavioral activation therapy focusing on meaningful and enjoyable, physical, cognitive and social activities has shown positive effects on quality of life and activity level as well as long-term benefits on cognition and daily functioning in patients with MCI and mild dementia. In addition, effects on neuropsychiatric symptoms such as depression are reasonable as behavioral activation therapy has strong and consistent effects on patients with depression. However, effects of a highly scalable, digital version of behavioral activation therapy in patients with MCI or mild dementia are not proven so far. Therefore, this study primarily aims to explore effects of the digital health app MindAhead Active in adults with MCI or mild dementia in a pilot study.

The primary objective of this study is to explore effect sizes in different outcomes (primary outcomes: quality of life, overall activity level) that will be used to calculate the sample size of a larger trial. The secondary objective is the validation of instruments. The investigators aim to validate three questionnaires that may depict outcomes of the full-scale study in case of success.

Further objectives are to assess feasibility regarding the study (recruitment of eligible subjects, online assessment, study completion/dropout rates), and the intervention (app installation, usage and intervention adherence/completion) as well as to confirm findings from previously conducted studies on face-to-face behavioral activation therapy reporting no safety issues and no increase in adverse events in contrast to a control group. This trial is a monocentric, randomized controlled, assessor-blinded superiority trial with two parallel groups.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cognitive impairment in MCI stage (ICD-10 codes: F06.7, F07.8) or mild dementia stage (ICD-10: F00.-*, F01.-, F03) due to all etiologies apart from etiologies described in F02.- (Pick's disease, Parkinson's disease, multiple sclerosis, Huntington's disease, HIV, Lewy body disease). Hence, etiologies of MCI and mild dementia include

  * Alzheimer's disease (e.g., F00.-*)
  * Vascular disease (e.g., F01.-) (exception in case of stroke: event occurred > 12 months ago without ongoing spontaneous remission)
  * Mixed diseases
  * Unclear etiologies
* MCI or mild dementia diagnosis assigned within the last 12 months by a neurologist or psychiatrist from our cooperation partners that fulfil adequate diagnosis procedures such as neuropsychological assessment, brain imaging, self- and/or third-party medical history interview, and potentially cerebrospinal fluid, positron emission tomography, or electrophysiological measures
* MCI or mild dementia diagnosis confirmed by a treating physician
* MMSE ≥ 24 or MoCA ≥ 18 (last date of assessment is decisive; needs to be within the last 12 months)
* Sufficient physical fitness to engage in physical activities (e.g., walking or cycling) as confirmed by a treating physician
* Age ≥ 50
* German language skills sufficient to understand German instructions of study assessments and of the intervention
* Ability and sufficient vision to operate a smartphone

Exclusion Criteria:

* possibly moderate or severe cognitive impairment (moderate or severe dementia), indicated by MMSE < 24 or MoCA < 18 (last date of assessment is decisive; needs to be within the last 12 months)
* Specific brain injury events within the last 12 months or with ongoing spontaneous remission due to

  * Stroke (ischemic, hemorrhagic)
  * Traumatic brain injury
* Specific etiologies of MCI or mild dementia (F02.-) that show a variable course or a fast progression including

  * Multiple sclerosis
  * Parkinson's disease
  * Pick's disease / Frontotemporal lobar degeneration
  * Lewy body disease
  * Brain tumors
  * Autosomal dominant form of Alzheimer's disease with early first manifestation
  * Creutzfeldt-Jakob disease
* German language restrictions or visual restrictions which prevent from understanding written German instructions of assessment or intervention procedures (e.g. severe aphasia, lack of sufficient German language skills, severe non-corrected visual impairment)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-12-21 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Overall Quality of Life | 3 months
  Change in quality of life (total score of generic and disorder-specific quality of life) from baseline to 3-month follow-up. Overall quality of life will be measured with a composite score of all items of the World Health Organization WHOQOL-BREF quality of life assessment and the Dementia Quality of Life (DEMQOL). All items will be transformed to a scale ranging from 0 to 100 and subsequently averaged. Higher scores indicate a higher quality of life.
Activity Level | 3 months
  Change in activity level (total score of social, physical and cognitive activity level) from baseline to 3-month follow-up. Overall activity level will be measured with the Community Healthy Activities Model Program for Seniors (CHAMPS) German version. The CHAMPS assesses frequency and duration of 41 physical, cognitive, and social activities of a typical week within the last 4 weeks. As measure for activity level, we assess the total hours spend per week covering all performed 41 activities, by adding up the data on activity duration (as described by Poelke, et al., 2016, International Psychogeriatrics). Therefore, the duration scale for each item is transformed as described in the original work by Stewart et al. (2001, Medicine and Science in Sports and Exercise), with category 1 = 0.5 hours, 2 = 1.75 hours, 3 = 3.75 hours, 4 = 5.75 hours, 5 = 7.75 hours, and 6 = 9.75 hours. The composite score can range from 0 to 399.75 hours per week.

SECONDARY OUTCOMES:
Disorder-specific quality of life | 3 months
  Change in disorder-specific quality of life from baseline to 3-month follow-up. Disorder-specific quality of life will be measured with the Dementia Quality of Life (DEMQOL) questionnaire. The DEMQOL contains 29 items with one overall quality of life item as well as 28 specific items covering positive and negative emotions, cognition and acitivities of daily living. For the total score the 28 specific items are used (scores ranging from 28 to 112, with higher scores indicating higher quality of life).
Generic quality of life - composite score | 3 months
  Change in generic quality of life from baseline to 3-month follow-up. Generic quality of life - composite score will be measured with the World Health Organization WHOQOL-BREF quality of life assessment. The WHOQOL-BREF total score is composed by the 26 items of all 4 WHOQOL-BREF subdomains (raw scores ranging from 26 to 130 are transformed to range from 0 to 100, with a higher score indicating higher quallity of life).
Generic quality of life - physical health subscale | 3 months
  Change from baseline to 3-month follow-up. Generic quality of life - physical health will be measured with the World Health Organization WHOQOL-BREF quality of life assessment - physical health subscale with 7 items (raw scores ranging from 7 to 35 are transformed to range from 0 to 100, with a higher score indicating higher physical health).
Generic quality of life - psychological health subscale | 3 months
  Change from baseline to 3-month follow-up. Generic quality of life - psychological health will be measured with the World Health Organization WHOQOL-BREF quality of life assessment - psychological health subscale with 6 items (raw scores ranging from 6 to 30 are transformed to range from 0 to 100, with a higher score indicating higher psychological health).
Generic quality of life - social relationships subscale | 3 months
  Change from baseline to 3-month follow-up. Generic quality of life - social relationships will be measured with the World Health Organization WHOQOL-BREF quality of life assessment - social relationships subscale with 3 items (raw scores ranging from 3 to 15 are transformed to range from 0 to 100, with a higher score indicating higher quality of social relationships).
Generic quality of life - environment subscale | 3 months
  Change from baseline to 3-month follow-up. Generic quality of life - environment will be measured with the World Health Organization WHOQOL-BREF quality of life assessment - environment subscale with 8 items (raw scores ranging from 8 to 40 are transformed to range from 0 to 100, with a higher score indicating higher environmental quality of life).
Generic quality of life - global subscale | 3 months
  Change from baseline to 3-month follow-up. Generic quality of life - environment will be measured with the World Health Organization WHOQOL-BREF quality of life assessment - global subscale with 2 items (raw scores ranging from 2 to 10 are transformed to range from 0 to 100, with a higher score indicating higher global quality of life).
Cognitive activity level | 3 months
  Change in cognitive activity level from baseline to 3-month follow-up. Cognitive activity levels will be measured with CHAMPS.
  The activities will be categorized to the three domains (physical, cognitive, and social activity level as described in Küster et al., 2016, BMC Psychiatry). The following activities are included in the cognitive domain: single-domain activities: play muscial instruments; use a computer; read; do arts and crafts; and multidomain acitivities: play basketball, soccer or raquetball; play singles tennis; play doubles tennis; dance; play cards and board games; visit family or friends; do volunteer work; attend club meetings; attend cultural meetings; do yoga or Tai Chi.
  The cognitive activity level domain score is then built as described in Poelke, et al. (2016, International Psychogeriatrics).
Physical activity level | 3 months
  Change in physical activity level from baseline to 3-month follow-up. Physical activity levels will be measured with the CHAMPS.
  The activities will be categorized to the three domains (physical, cognitive, and social activity level as described in Küster et al., 2016, BMC Psychiatry). The following activities are included in the physical domain: single-domain activities: jog or run; swim moderately or fast; skate; use an aerobic machine; do moderate/heavy strength training; walk uphill or hike; do heavy gardening; do water exercise; bicycle; do heavy work around the house; and multidomain acitivities: play basketball, soccer or raquetball; play singles tennis; play doubles tennis; dance; do yoga or Ta Chi; do aerobic; play golf with carrying equipment.
  The physical activity level domain score is then built as described in Poelke, et al. (2016, International Psychogeriatrics).
Social activity level | 3 months
  Change in social activity level from baseline to 3-month follow-up. Social activity levels will be measured with the CHAMPS.
  The activities will be categorized to the three domains (physical, cognitive, and social activity level as described in Küster et al., 2016, BMC Psychiatry). The following activities are included in the social domain: single-domain activities: go to the senior center; attend curch activities; and multidomain acitivities: play basketball, soccer or raquetball; play singles tennis; play doubles tennis; dance; play cards and board games; visit family or friends; do volunteer work; attend club meetings; attend cultural events; do aerobic; play golf with carrying equipment.
  The social activity level domain score is then built as described in Poelke, et al. (2016, International Psychogeriatrics).
Depressive symptoms | 3 months
  Change in depressive symptoms from baseline to 3-month follow-up. Depressive symptoms will be measured with the Geriatric Depression Scale 30 (GDS-30). The GDS contains 30 items (scores range from 0 to 30 with higher scores indicating greater depression).
Subjective cognitive symptoms - everyday memory | 3 months
  Change in subjective cognitive symptoms from baseline to 3-month follow-up. Subjective cognitive symptoms will be measured with the Everyday Memory Survey (EMS). The EMS contains 25 items of which 23 items are included into the total score (scores range from 0 to 92, with higher scores indicating greater subjective cognitive symptoms - everyday memory).
Subjective cognitive symptoms - global cognition | 3 months
  Change in subjective cognitive symptoms from baseline to 3-month follow-up. Subjective cognitive symptoms - global cognition will be measured with a new German version of the British Columbia - Cognitive Complaints Inventory (BC-CCI). The BC-CCI contains 6 items (scores range from 0 to 18, with higher scores indication greater subjective cognitive complaints).
Chronic disease-specific quality of life | 3 months
  Change in chronic disease-specific quality of life from baseline to 3-month follow-up, measured with the German Quality of Life Scale (QOLS-G). The QOLS-G contains 16 items which are summed up to a sum score (scores range from 16 to 112, with higher scores indicating higher level of satisfaction).
Neurocognitive disorder-specific quality of life | 3 months
  Change in neurocognitive disorder-specific quality of life from baseline to 3-month follow-up, measured with the newly developed Quality of Life-Neurocognitive Disorder (QoL-NCD), which is based on the Mild Cognitive Impairment Questionnaire and the Dementia Quality of Life (DEMQOL)-self report. The QoL-NCD contains 25 items, with a superordinate item on general quality of life and 6 items for each of the 4 domains: cognitive health, psychological health, activities of daily living, and social relationships. The total score includes all 25 items (range from 0 to 100 with higher scores indication higher quality of life).
Goal-oriented activity level | 3 months
  Change in goal-oriented activity level from baseline to 3-month follow-up. Goal-oriented activity level will be measured with the activation subscale of the Behavioral Activation for Depression Scale (BADS). The BADS Activation subscale contains 7 items (scores range from 0 to 42, with higher scores indicating a higher goal-oriented activity level).
Domain-specific activity level | 3 months
  Change in domain-specific activity level from baseline to 3-month follow-up. Domain-specific activity level will be measured with the newly developed Meaningful, Enjoyable, Physical, Social, and Cognitive Activity Scale (MEPSCAS). The MEPSCAS contains of 5 items, assessing physical, cognitive, social, enjoyable and meaningful activity on a 10-point rating scale from 1 ("not at all") to 10 ("extremely"). The domain-specific activity level composite scores will be built by averaging all available items, thus ranging from 1 to 10, with higher scores depicting higher domain-specific activity.

OTHER OUTCOMES:
Daily functioning | 3 months
  Change in daily functioning from baseline to 3-month follow-up. Daily functioning will be measured with the Bayer-Activities of Daily Living Scale (B-ADL). The B-ADL contains 25 items. The composite score depicts the mean scoring in all available items with a possible range from 1 to 10.
General patient satisfaction | 3 months
  General patient satisfaction from baseline to 3-month follow-up. General patient satisfaction will be measured with the patient satisfaction questionnaire (PSQ) - general satisfaction scale. The PSQ general satisfaction subscale contains 2 items (scores range from 1 to 5, higher scores depicting higher satisfaction).
Screening time | 3 months
  To assess feasibility of study procedures, the time required to screen one patient will be assessed.
Recruiting time | 3 months
  To assess feasibility of study procedures, the time required to recruit one patient will be assessed.
Inclusion rate | 3 months
  To assess feasibility of study procedures, the percentage of included patients to screened patients will be assessed.
Study completion rate | 3 months
  To assess feasibility of study procedures, the dropout rates (the percentage of patients completing the 3-month follow-up assessment) in expected primary outcomes will be assessed.
Intervention completion rate | 3 months
  To assess feasibility of and adherence to the intervention, the rate of participants who completed the intervention will be assessed. The intervention is defined to be completed, if at least 13 units, including repeated units, have been carried out (i.e., on average at least 1 unit per week).
Completed activity goals | 3 months
  To assess feasibility of and adherence to the intervention, the number of completed activity goals in the MindAhead Active app will be assessed for all participants of the intervention group.
App logins / accesses | 3 months
  To assess feasibility of and adherence to the intervention, the app usage is assessed by the average number the app has been accessed.
Scheduled activities | 3 months
  To assess feasibility of and adherence to the intervention, the average number of planned activity goals is obtained.
Major Adverse Events (MAE) | 3 months
  Number of predefined major adverse events: Number of falls, injuries, and hospitalizations will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Jens Wiltfang, Prof. Dr., Principal Investigator — University Medical Center Göttingen, Clinic for Psychiatry and Psychotherapy, Germany; Christine A.F. von Arnim, Prof. Dr., Principal Investigator — University Medical Center Göttingen, Clinic for Geriatrics, Germany
Locations (1):
- University Medical Center Göttingen, Göttingen, Germany

IPD SHARING:
Plan to Share IPD: Undecided